CLINICAL TRIAL: NCT01604538
Title: Italian Pulmonary Embolism Registry
Brief Title: Italian Pulmonary Embolism Registry - IPER
Acronym: IPER
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Cecilia Becattini, Dr, University Of Perugia
Other Study IDs: protocol_364
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with acute pulmonary embolism

SUMMARY:
RAZIONALE

Pulmonary embolism is a complex disease, with a highly variable clincal presentation. Diagnosis starts with clinical probability assessment mainly based on medical history and rapidly available clinical data. Pulmonary embolism can be managed by emergency department, cardiology, pneumology geriatrics or internal medicine physicians. Thus, initial clinical management can varies based on the attitude of the attending physician.

Diagnosis is a crucial point as it can influence short term mortality.

OBJECTIVE

The registry has 3 main objectives:

1. educational objective,
2. improvement in the knowledge of epidemiology, management and outcome of acute pulmonary embolism in Italy
3. scientific objective

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with acute pulmonary embolism

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Franco Casazza, MD, Study Chair — San Carlo Borromeo hospital, Milan, Italy

REFERENCES:
- [Derived] Zuin M, Bilato C, Enea I, Bongarzoni A, Casazza F, Roncon L, Becattini C. An exploratory model for short-term risk stratification in intermediate-high-risk pulmonary embolism running head: The STAMP score. Eur J Intern Med. 2026 Feb;144:106484. doi: 10.1016/j.ejim.2025.106484. Epub 2025 Aug 20. PMID 40841246
- [Derived] Zuin M, Piazza G, Rigatelli G, Bongarzoni A, Enea I, Casazza F, Picariello C, Bilato C, Roncon L. Clinical phenotypes and risk of early hemodynamic deterioration in intermediate-high-risk patients with acute pulmonary embolism. Thromb Res. 2025 Aug;252:109380. doi: 10.1016/j.thromres.2025.109380. Epub 2025 Jun 10. PMID 40505225
- [Derived] Zuin M, Rigatelli G, Bilato C, Bongarzoni A, Zonzin P, Casazza F, Roncon L. Risk of early clinical deterioration and 30-day mortality in pulmonary embolism intermediate-high-risk patients with patent foramen ovale. Intern Emerg Med. 2024 Sep;19(6):1637-1644. doi: 10.1007/s11739-024-03657-w. Epub 2024 May 31. PMID 38822190
- [Derived] Zuin M, Piazza G, Rigatelli G, Bilato C, Bongarzoni A, Henkin S, Zonzin P, Casazza F, Roncon L. Prognostic Role of Tricuspid Annular Plane Systolic Excursion to Systolic Pulmonary Artery Pressure Ratio for the Identification of Early Clinical Deterioration in Intermediate-High-Risk Pulmonary Embolism Patients. Am J Cardiol. 2024 Mar 1;214:40-46. doi: 10.1016/j.amjcard.2023.12.053. Epub 2024 Jan 11. PMID 38218392
- [Derived] Zuin M, Bilato C, Bongarzoni A, Zonzin P, Casazza F, Roncon L. Prognostic impact of the e-TAPSE ratio in intermediate-high risk pulmonary embolism patients. Int J Cardiovasc Imaging. 2024 Mar;40(3):467-476. doi: 10.1007/s10554-023-03010-w. Epub 2023 Nov 30. PMID 38032504
- [Derived] Zuin M, Rigatelli G, Bongarzoni A, Enea I, Bilato C, Zonzin P, Casazza F, Roncon L. Mean arterial pressure predicts 48 h clinical deterioration in intermediate-high risk patients with acute pulmonary embolism. Eur Heart J Acute Cardiovasc Care. 2023 Feb 9;12(2):80-86. doi: 10.1093/ehjacc/zuac169. PMID 36580441
- [Derived] Zuin M, Bilato C, Bongarzoni A, Zonzin P, Casazza F, Rigatelli G, Roncon L. Impact of clinical profile at admission on the outcomes in patients hospitalized for acute pulmonary embolism: data from the IPER Registry. J Thromb Thrombolysis. 2023 Jan;55(1):166-174. doi: 10.1007/s11239-022-02726-1. Epub 2022 Nov 9. PMID 36350468
- [Derived] Becattini C, Casazza F, Forgione C, Porro F, Fadin BM, Stucchi A, Lignani A, Conte L, Imperadore F, Bongarzoni A, Agnelli G. Acute pulmonary embolism: external validation of an integrated risk stratification model. Chest. 2013 Nov;144(5):1539-1545. doi: 10.1378/chest.12-2938. PMID 23764909